CLINICAL TRIAL: NCT05587465
Title: Evaluation of Safety and Effectiveness of Lobster Dynamic Interspinous Spacer in Lumbar Spinal Stenosis: A Single Arm, Prospective, Mutli-Center Study
Brief Title: Evaluation of Safety and Effectiveness of Lobster Dynamic Interspinous Spacer in Lumbar Spinal Stenosis
Acronym: LB2CT01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diametros Medical srl (Industry)
Collaborators: MCRA (Industry); Sciently di Omar Sabry (Unknown); Medical Consulting srl (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 446/2022/CE
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Spinal Lumbar Stenosis; Claudication, Intermittent
Keywords: Radiology; Interspinous Spacer; Interventional Radiology; Neurosurgery; Vertebral surgery; Pain management; Neurogenic intermittent claudicatio; Degenerative disc disease; Percutaneous operating technique
MeSH Terms: conditions — Intermittent Claudication; Agnosia; Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: single arm, prospective, multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Lobster device implantation
  Interventions: Device: Lobster Device

INTERVENTIONS:
Device: Lobster Device — The intervention is performed percutaneously using the dedicated instrument set.
  Other Names: Interspinous Spacer implantation

SUMMARY:
The aim of this study is to demonstrate the safety and effectiveness of the Lobster interspinous spacer device for the treatment of Lumbar Spinal Stenosis in comparison to an SSED-based performance goal.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, patients with Lumbar Spinal Stenosis matching inclusion and exclusion criteria giving written informed consent will undergo Lobster device implantation and followed-up for 2 years for radiological and clinical assessment in a single-arm, prospective, multicentric clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 45 years of age.
2. Persistent leg/buttock/groin pain, with or without back pain, that is relieved by flexion activities (example: sitting or bending over a shopping cart).
3. Subjects who have been symptomatic and undergoing conservative care treatment for at least 6 months.
4. Diagnosis of degenerative spinal stenosis of the lumbar spine, defined as the narrowing of the midline sagittal spinal canal (central) and/or narrowing between the facet superior articulating process (SAP), the posterior vertebral margin (lateral recess), and the nerve root canal (foraminal).
5. Radiographic confirmation of at least moderate spinal stenosis which narrows the central, lateral, or foraminal spinal canal at one or two contiguous levels from L1-L5. Moderate spinal stenosis is defined as 25% to 50% reduction in lateral/central foramen compared to the adjacent levels, with radiographic confirmation of any one of the following:

   1. Evidence of thecal sac and/or cauda equina compression.
   2. Evidence of nerve root impingement (displacement or compression) by either osseous or non-osseous elements.
   3. Evidence of hypertrophic facets with canal encroachment.

   Note: All imaging studies used to confirm LSS are to be completed within 3 months prior to enrollment. Radiographic (imaging) confirmation of LSS included MRI and/or CT. In the case of a transitional L5/L6 segment with a sufficiently prominent L6 spinous process, these subjects may be included by a deviation request from the applicant.
6. Must present with moderately impaired Physical Function (PF) defined as a score of > 2.0 of the Zurich Claudication Questionnaire (ZCQ).
7. Must be able to sit for 50 minutes without pain and to walk 15 meters (50 feet) or more .
8. Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
9. Subjects, who, in the opinion of the Clinical Investigator, are able to understand this clinical investigation, cooperate with the investigational procedures and are willing to return for all the required post-treatment follow-ups.

Exclusion Criteria:

1. Axial back pain only.
2. Fixed motor deficit.
3. Diagnosis of lumbar spinal stenosis which requires any direct neural decompression or surgical intervention other than those required to implant the control or investigational device.
4. Unremitting pain in any spinal position.
5. Significant peripheral neuropathy or acute denervation secondary to radiculopathy.
6. Lumbar spinal stenosis at more than two levels determined pre-operatively to require surgical intervention.
7. Significant instability of the lumbar spine as defined by ≥ 3mm translation or ≥ 5° angulation.
8. Sustained pathologic fractures of the vertebrae or multiple fractures of the vertebrae and/or hips.
9. Spondylolisthesis or degenerative spondylolisthesis greater than grade 1 (on a scale of 1-4).
10. Spondylolysis (pars fracture).
11. Degenerative lumbar scoliosis with a Cobb angle of > 10° at treatment level.
12. Osteopenia or osteoporosis. To confirm eligibility, at the Clinical Investigator's discretion, the following subjects may have a DEXA scan performed:

    i. Women 65 or older ii. Postmenopausal women < age 65 iii. Subjects with major risk factors for or diagnosed with osteoporosis or osteopenia iv. If DEXA is required, exclusion is defined as a DEXA bone density measurement T score ≤ -2.5
13. Morbid obesity, defined as Body Mass Index (BMI) greater than 40kg/m2.
14. Insulin-dependent diabetes mellitus.
15. Significant peripheral vascular disease (diminished dorsalis pedis or tibial pulses).
16. Prior surgery of the lumbar spine.
17. Cauda equina syndrome (defined as neural compression causing neurogenic bowel or bladder dysfunction).
18. Infection in the disc or spine, past or present.
19. Evidence of active (systemic or local) infection at time of surgery.
20. Active systemic disease such as AIDS, HIV, hepatitis, etc.
21. Paget's disease at involved segment or metastasis to the vertebra, osteomalacia, or other metabolic bone disease.
22. Currently undergoing immunosuppressive therapy or long-term steroid use.
23. Known allergy to titanium or titanium alloys.
24. Tumor in the spine or a malignant tumor except for basal cell carcinoma 25. Known or suspected history of alcohol and/or drug abuse.
25. Prisoner or transient.
26. Life expectancy less than two years.
27. Angina, active rheumatoid arthritis, or any other systemic disease that would affect the subject's welfare or outcome of the clinical investigation.
28. Any significant mental illness (e.g., major depression, schizophrenia, bipolar disorder, etc.) that could impair the consent process or ability to complete subject self-report questionnaires.
29. Involved in pending litigation of the spine or worker's compensation related to the back.
30. Enrolled in the treatment phase of another drug or device clinical investigation (currently or within past 30 days).
31. Congenital defect of the spine.
32. Pregnant or lactating.
33. Any further contraindications and limitations of the device as described in the instructions for use (IFU).

Subjects who meet any of the following criteria will be excluded from participating in this study:

1. Axial back pain only.
2. Fixed motor deficit.
3. Diagnosis of lumbar spinal stenosis which requires any direct neural decompression or surgical intervention other than those required to implant the control or investigational device.
4. Unremitting pain in any spinal position.
5. Significant peripheral neuropathy or acute denervation secondary to radiculopathy.
6. Lumbar spinal stenosis at more than two levels determined pre-operatively to require surgical intervention.
7. Significant instability of the lumbar spine as defined by ≥ 3mm translation or ≥ 5° angulation.
8. Sustained pathologic fractures of the vertebrae or multiple fractures of the vertebrae and/or hips.
9. Spondylolisthesis or degenerative spondylolisthesis greater than grade 1 (on a scale of 1-4).
10. Spondylolysis (pars fracture).
11. Degenerative lumbar scoliosis with a Cobb angle of > 10° at treatment level.
12. Osteopenia or osteoporosis. To confirm eligibility, at the Clinical Investigator's discretion, the following subjects may have a DEXA scan performed:

    i. Women 65 or older ii. Postmenopausal women < age 65 iii. Subjects with major risk factors for or diagnosed with osteoporosis or osteopenia iv. If DEXA is required, exclusion is defined as a DEXA bone density measurement T score ≤ -2.5
13. Morbid obesity, defined as Body Mass Index (BMI) greater than 40kg/m2.
14. Insulin-dependent diabetes mellitus.
15. Significant peripheral vascular disease (diminished dorsalis pedis or tibial pulses).
16. Prior surgery of the lumbar spine.
17. Cauda equina syndrome (defined as neural compression causing neurogenic bowel or bladder dysfunction).
18. Infection in the disc or spine, past or present.
19. Evidence of active (systemic or local) infection at time of surgery.
20. Active systemic disease such as AIDS, HIV, hepatitis, etc.
21. Paget's disease at involved segment or metastasis to the vertebra, osteomalacia, or other metabolic bone disease.
22. Currently undergoing immunosuppressive therapy or long-term steroid use.
23. Known allergy to titanium or titanium alloys.
24. Tumor in the spine or a malignant tumor except for basal cell carcinoma 25. Known or suspected history of alcohol and/or drug abuse.
25. Prisoner or transient.
26. Life expectancy less than two years.
27. Angina, active rheumatoid arthritis, or any other systemic disease that would affect the subject's welfare or outcome of the clinical investigation.
28. Any significant mental illness (e.g., major depression, schizophrenia, bipolar disorder, etc.) that could impair the consent process or ability to complete subject self-report questionnaires.
29. Involved in pending litigation of the spine or worker's compensation related to the back.
30. Enrolled in the treatment phase of another drug or device clinical investigation (currently or within past 30 days).
31. Congenital defect of the spine.
32. Pregnant or lactating.
33. Any further contraindications and limitations of the device as described in the instructions for use (IFU).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the Lobster device in comparison to an SSED-based performance goal (PG) | 12 months
  Efficacy success will be evaluated as a two-prong composite endpoint:
  * ZCQ Responder (at least two of the three ZCQ domains)
    * ≥0.5 point improvement in physical function
    * ≥0.5 point improvement in symptom severity
    * Mean satisfaction ≤2.5 points
  * No secondary surgical intervention (SSI) including re-operations, revision, removals or supplemental fixation or clinical significant confounding treatments (i.e., epidural steroid injections at the index level, spinal cord stimulators or rhizotomies) through 12 months
Safety of the Lobster device in comparison to an SSED-based performance goal (PG) | 12 months
  Safety success will be evaluated using precision-based statistics to characterize the incidence of major device- or procedure-related complications, including:
  * Device integrity failure (dislodgement, migration, or deformation)
  * New or persistent worsened neurological deficit at the index level
  * Spinous process fractures
  * Deep infection, death, or other permanent device attributed disability

SECONDARY OUTCOMES:
Oswestry disability index (ODI) | Pre-treatment, 6 weeks, 3 months, 6 months, 12 months, 24 months
  Oswestry disability index. Patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain.
  Min. value 0 (better outcome) Max. value 100 (worst outcome)
Visual Analogue Scale (VAS) | Pre-treatment, 6 weeks, 3 months, 6 months, 12 months, 24 months
  VAS (Pain regarding Back and Leg)
  Min. value 0 (better outcome) Max. value 10 (worst outcome)
Short Form SF-12 | Pre-treatment, 6 weeks, 3 months, 6 months, 12 months, 24 months
  SF-12 Short Form Survey (Physical Function and Mental Health). The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  Min. value 0 (worst outcome) Max. value 100 (better outcome)
Zurich Claudication Questionnaire (ZCQ) | Pre-treatment, 6 weeks, 3 months, 6 months, 12 months, 24 months
  The questionnaire consists of three domains and uses a Likert-type scale. It includes 7 items for symptom severity with scores of 1 to 5, 5 items for functional disability with scores of 1 to 4, and 6 items for treatment satisfaction with score of 1 to 4. Higher scores indicate more severe LSS.
Number of participants with abnormal Neurological examination findings | Pre-treatment, 6 weeks, 3 months, 6 months, 12 months, 24 months
  Neurological examination to assess and identify any abnormalities that affect function and activities of daily living. Electromyography is performed at the discretion of the investigator.
Radiological status | Pre-treatment, 6 weeks, 3 months, 6 months, 12 months, 24 months
  An independent radiographic core laboratory will be used to provide an unbiased assessment of all x-rays and CT scans (pre-procedure through last follow-up assessment). All images will be evaluated in accordance with the Image Review Charter which is provided to the sites.
  Radiographic evaluations include:
  * Angular Range of Motion
  * Translational Motion
  * Device Condition
  * Device Migration
  * Device Dislodgement
  * Bone-Implant Interface Changes
  * Exuberant Bone Formation

CONTACTS AND LOCATIONS:
Locations (1):
- SS. Trinità - Reparto di Radiologia, Cagliari, Sardinia, Italy

DOCUMENTS (1):
  • Study Protocol (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT05587465/Prot_000.pdf